CLINICAL TRIAL: NCT06854666
Title: Clinical and Morphological Evaluation Following Treatment of Lateral Epicondylar Tendinopathy with PRP or L-PRP,saline- Prospective Randomized Double Blinded Controlled Trial
Brief Title: Leukocyte-Poor Platelet-Rich Plasma Reduces Pain Symptoms in the Treatment of the Lateral Epicondylitis
Acronym: LET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehasport Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSC_JWAL_2024_V1; Secec grant 2017 (Other Grant/Funding Number: European Society for Surgery of the Shoulder and the Elbow)
Record Dates: First submitted 2025-01-13; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Tennis Elbow; Lateral Epicondylitis; Lateral Epicondylitis (tennis Elbow); PRP Injection; PRP and Physiotherapy
Keywords: tennis elbow; prp
MeSH Terms: conditions — Tennis Elbow; Insomnia, Fatal Familial

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standardized PRP Injection (Active Comparator): A standardized PRP preparation protocol (without commercial kits) is used, ensuring consistency in platelet concentration.
  Preparation Process:
  Blood Collection: 30 ml of venous blood drawn from each patient Centrifugation: 7 minutes at 2,054 g using MPV-223e centrifuge Separation: Blood fractionated into erythrocytes, leukocytes, PRP, and platelet-poor plasma PRP Isolation: Pure PRP extracted for injection Injection Procedure: 2 ml of PRP injected into the tendon pain area, with 1 ml retained for laboratory analysis
  Interventions: Other: effectiveness of platelet-rich plasma (PRP) in treating lateral epicondylar tendinopathy (LET)
- Standardized leukocyte-rich PRP (L-PRP) (Active Comparator): A standardized leukocyte-rich PRP (L-PRP) preparation protocol (without commercial kits) is used to ensure consistency in platelet and leukocyte concentrations.
  Preparation Process:
  Blood Collection: 30 ml of venous blood drawn from each patient Centrifugation: 7 minutes at 2,054 g using MPV-223e centrifuge Separation: Blood fractionated into erythrocytes, leukocytes, PRP, and platelet-poor plasma L-PRP Isolation: Leukocyte-rich PRP extracted for injection Injection Procedure: 2 ml of L-PRP injected into the tendon pain area, with 1 ml retained for laboratory analysis
  Interventions: Other: effectiveness of platelet-rich plasma (PRP) in treating lateral epicondylar tendinopathy (LET)
- Saline Injection (Placebo Control) (Active Comparator): A placebo control group receiving a standardized saline injection to evaluate the efficacy of PRP and L-PRP treatments.
  Procedure:
  Injection of 2 ml of sterile saline into the tendon pain area, following the same protocol as the PRP and L-PRP groups.
  Interventions: Other: effectiveness of platelet-rich plasma (PRP) in treating lateral epicondylar tendinopathy (LET)

INTERVENTIONS:
Other: effectiveness of platelet-rich plasma (PRP) in treating lateral epicondylar tendinopathy (LET) — The intervention involves the administration of PRP (platelet-rich plasma), L-PRP (leukocyte-rich platelet-rich plasma), and saline according to a protocol developed for patients with lateral epicondylitis (EPi lat). The intervention includes specific parameters such as centrifugation speed and dual injection to the painful site, which is repeated after one week.
  Following the procedure, treatment continues with a rehabilitation program, including the use of an orthosis. The orthosis serves as support during the recovery process after the injection. The rehabilitation program and the use of the orthosis aim to improve joint function and reduce pain, supporting tissue healing and regeneration.

SUMMARY:
Lateral epicondylar tendinopathy (LET), or tennis elbow, is a degenerative condition affecting the forearm's extensor tendons. It commonly leads to pain, reduced grip strength, and impaired function, particularly in individuals performing repetitive wrist and forearm movements. Standard treatments, including physiotherapy, braces, and anti-inflammatory medications, provide relief but do not always lead to full recovery. Platelet-rich plasma (PRP) has gained interest as a regenerative therapy with the potential to enhance tendon healing and improve clinical outcomes.

This randomized, double-blind, placebo-controlled trial aims to evaluate PRP's effectiveness in treating LET, comparing it to leukocyte-rich PRP (L-PRP) and saline (placebo). Additionally, it assesses the composition of PRP and its role in tendon regeneration.

The study will enroll 80 patients diagnosed with LET, meeting predefined clinical criteria. Participants will be randomized into three groups (PRP, L-PRP, saline) and receive two injections (day 0 and day 7). PRP will be prepared using a standardized protocol to ensure consistency.

Patients will undergo clinical evaluations (VAS, Mayo Elbow Score, SECEC Elbow Score), grip strength testing, and MRI scans at baseline and 24 weeks post-treatment. The PRP composition will be analyzed in a laboratory. Follow-ups will be conducted at 12, 24, and 54 weeks to monitor pain reduction, functional improvement, and tendon healing.

This study will provide critical insights into PRP's therapeutic potential, helping refine treatment approaches for LET and improve patient outcomes.

DETAILED DESCRIPTION:
Detailed Description

Study Rationale

Lateral epicondylar tendinopathy (LET), commonly referred to as tennis elbow, is a chronic degenerative condition affecting the common extensor tendon (CET) at the lateral epicondyle of the humerus. It is commonly observed in individuals engaged in repetitive wrist and forearm movements, such as athletes, manual laborers, and office workers. The primary pathological mechanism involves microtears leading to pain, reduced grip strength, and impaired function.

Conservative treatments, including physiotherapy, nonsteroidal anti-inflammatory drugs (NSAIDs), corticosteroid injections, and bracing, often provide temporary symptom relief but do not facilitate tendon regeneration. Corticosteroid injections may offer short-term pain relief but have been associated with tendon degeneration and higher recurrence rates. Given the limitations of these treatments, platelet-rich plasma (PRP) has emerged as a promising biological therapy due to its high concentration of growth factors that promote tissue healing, angiogenesis, and anti-inflammatory effects.

However, the optimal formulation of PRP remains controversial. Some studies suggest that leukocyte-rich PRP (L-PRP) may enhance the inflammatory response and accelerate healing, while others indicate that leukocyte-poor PRP (LP-PRP) may have superior effects by reducing excessive inflammation. The cellular composition of PRP is not standardized across clinical studies, leading to variability in treatment outcomes. This study seeks to clarify the role of PRP in LET treatment, determine whether L-PRP offers superior benefits, and evaluate its effects on pain relief, functional recovery, and tendon healing over time.

Study Design and Methodology

This is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the efficacy of PRP and L-PRP, saline compared to saline injections in treating LET. The study will enroll 80 symptomatic patients diagnosed with LET based on clinical criteria. Patients will be randomly assigned to one of the three treatment groups:

PRP Group (n=20): Standard platelet-rich plasma injection

L-PRP Group (n=20): Leukocyte-rich platelet-rich plasma injection

Saline Group (Control) (n=20): Placebo (saline) injection

Both PRP and L-PRP will be prepared using a standardized, non-commercial protocol to ensure consistency in cellular composition. Blinding procedures will ensure that neither the patients nor the evaluating clinicians know which treatment is administered.

Patient Selection Criteria

Inclusion Criteria:

Age 18-65 years

Diagnosed with chronic lateral epicondylitis (duration >6 months)

Positive clinical tests: pain on resisted wrist extension and decreased grip strength

Written informed consent

Exclusion Criteria:

Previous elbow surgery or PRP treatment

Corticosteroid injections within the past 3 months

Systemic inflammatory or autoimmune diseases

Pregnancy or breastfeeding

Neurological conditions affecting upper limb function

PIN syndrome

Treatment Protocol

Pre-Treatment Evaluation:

All patients will undergo:

Clinical assessment of pain and function

VAS and Oxford Elbow Score questionnaires

Grip strength testing using BTE

MRI imaging of the affected elbow (baseline)

Injection Procedure:

Blood Collection: 30 ml of venous blood will be drawn from each patient

Centrifugation: Blood will be centrifuged at 2054 g for 7 minutes to separate PRP fractions

PRP/L-PRP Preparation: The appropriate PRP fraction will be extracted (with or without leukocytes)

Injection: 2 ml of PRP or L-PRP will be injected into the CET, with 1 ml retained for laboratory analysis

Control Group: Patients will receive an equivalent saline injection following the same procedure

Post-Treatment Rehabilitation:

Guided physiotherapy program focusing on eccentric strengthening

Use of elbow braces during daily activities

Activity modification guidelines

Outcome Measures and Follow-Up

Primary Outcome:

Pain reduction measured by VAS score

Secondary Outcomes:

Functional improvement assessed using Oxford Elbow Score

Grip strength recovery using a digital dynamometer BTE Structural tendon healing assessed via MRI at baseline and 24 weeks post-treatment

Follow-Up Schedule:

Week 0: Baseline assessments and first injection

Week 1: Second injection

Week 12: First follow-up visit (VAS, Oxford Elbow Score, grip strength)

Week 24: Second follow-up visit (MRI assessment, VAS, Oxford Elbow Score, grip strength)

Week 54: Final follow-up visit (long-term clinical evaluation, VAS, Oxford Elbow Score, grip strength)

Laboratory Analysis

PRP samples will be analyzed for platelet concentration, leukocyte content, and growth factor levels

Comparative analysis between PRP and L-PRP to correlate biological composition with clinical outcomes

Expected Impact and Clinical Relevance

This study aims to establish a standardized PRP protocol for LET treatment and determine whether PRP offers superior benefits compared to conventional approaches. The results will provide:

High-quality evidence for clinicians regarding PRP effectiveness

Guidance on PRP formulation (leukocyte-rich vs. leukocyte-poor)

Objective MRI data to track structural healing of the common extensor tendon

Improved treatment strategies to enhance patient recovery and reduce recurrence rates

By correlating PRP composition with clinical and imaging outcomes, this trial will help refine biologic treatment strategies for chronic tendinopathies, ultimately improving evidence-based management of LET.

ELIGIBILITY:
Inclusion Criteria:

* first-time diagnosis of chronic lateral epicondylitis with a duration of at least 1 month, age of 18 years or more, and signed informed consent to participate in the study

Exclusion Criteria:

* pregnancy, any previous treatment for the condition (including injections around the elbow, rehabilitation, or use of orthoses), previous surgical treatment of the elbow, other painful elbow conditions, co-existing upper limb and/or neck pain, prior elbow trauma or arthritic changes, posterior interosseous nerve (PIN) neuropathy, and systemic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Improvement in Pain (VAS Score) | 12 months
  Description: This study aims to evaluate whether PRP reduces pain in patients with lateral epicondylar tendinopathy (LET).
  Assessment Tool: Visual Analog Scale (VAS) Scale: 0 to 10 (0 = no pain, 10 = worst possible pain) Higher scores indicate worse pain outcomes. Time Frame: 12 months
Grip Strength | 12 months
  Grip Strength: The study includes grip strength testing with isometric grip strenght measure BTE, which is a primary measure of functional improvement following treatment.
Improvement in Functional Outcomes (Oxford Elbow Score - OES) | 12 months
  Description: This study will assess whether PRP improves elbow function and daily activity performance in LET patients.
  Assessment Tool: Oxford Elbow Score (OES) Scale: 0 to 48 (0 = worst function/pain, 48 = best function/pain) Higher scores indicate better functional outcomes.

OTHER OUTCOMES:
Healing Process of Tendons | 12 months
  Healing Process of Tendons: The healing progress of the repaired tendons will be monitored using MRI imaging at before and after 24 weeks post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Walecka, MD, PhD, Principal Investigator — Rehasport Clinic; Przemyslaw Lubiatowski, MD, Phd,, Study Director — Rehasport Clinic
Locations (1):
- Rehasport, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kushida S, Kakudo N, Morimoto N, Hara T, Ogawa T, Mitsui T, Kusumoto K. Platelet and growth factor concentrations in activated platelet-rich plasma: a comparison of seven commercial separation systems. J Artif Organs. 2014 Jun;17(2):186-92. doi: 10.1007/s10047-014-0761-5. Epub 2014 Apr 20. PMID 24748436
- [Background] Dohan Ehrenfest DM, Rasmusson L, Albrektsson T. Classification of platelet concentrates: from pure platelet-rich plasma (P-PRP) to leucocyte- and platelet-rich fibrin (L-PRF). Trends Biotechnol. 2009 Mar;27(3):158-67. doi: 10.1016/j.tibtech.2008.11.009. Epub 2009 Jan 31. PMID 19187989
- [Background] Chaudhury S, de La Lama M, Adler RS, Gulotta LV, Skonieczki B, Chang A, Moley P, Cordasco F, Hannafin J, Fealy S. Platelet-rich plasma for the treatment of lateral epicondylitis: sonographic assessment of tendon morphology and vascularity (pilot study). Skeletal Radiol. 2013 Jan;42(1):91-7. doi: 10.1007/s00256-012-1518-y. Epub 2012 Sep 22. PMID 23001116
- [Background] Fulginiti VA. A new pertussis vaccine: hope for the future? J Infect Dis. 1983 Jul;148(1):146-7. doi: 10.1093/infdis/148.1.146. No abstract available. PMID 6350485
- [Background] Palacio EP, Schiavetti RR, Kanematsu M, Ikeda TM, Mizobuchi RR, Galbiatti JA. Effects of platelet-rich plasma on lateral epicondylitis of the elbow: prospective randomized controlled trial. Rev Bras Ortop. 2016 Jan 13;51(1):90-5. doi: 10.1016/j.rboe.2015.03.014. eCollection 2016 Jan-Feb. PMID 26962506
- [Background] Dronamraju KR. The origins of human gene mapping. With particular reference to the contributions of J. B. S. Haldane. Genomics. 1987 Nov;1(3):270-6. doi: 10.1016/0888-7543(87)90054-1. PMID 3328738
- [Background] Yadav R, Kothari SY, Borah D. Comparison of Local Injection of Platelet Rich Plasma and Corticosteroids in the Treatment of Lateral Epicondylitis of Humerus. J Clin Diagn Res. 2015 Jul;9(7):RC05-7. doi: 10.7860/JCDR/2015/14087.6213. Epub 2015 Jul 1. PMID 26393174
- [Background] Gautam VK, Verma S, Batra S, Bhatnagar N, Arora S. Platelet-rich plasma versus corticosteroid injection for recalcitrant lateral epicondylitis: clinical and ultrasonographic evaluation. J Orthop Surg (Hong Kong). 2015 Apr;23(1):1-5. doi: 10.1177/230949901502300101. PMID 25920633
- [Background] Italiano JE Jr, Richardson JL, Patel-Hett S, Battinelli E, Zaslavsky A, Short S, Ryeom S, Folkman J, Klement GL. Angiogenesis is regulated by a novel mechanism: pro- and antiangiogenic proteins are organized into separate platelet alpha granules and differentially released. Blood. 2008 Feb 1;111(3):1227-33. doi: 10.1182/blood-2007-09-113837. Epub 2007 Oct 25. PMID 17962514
- [Background] El-Sharkawy H, Kantarci A, Deady J, Hasturk H, Liu H, Alshahat M, Van Dyke TE. Platelet-rich plasma: growth factors and pro- and anti-inflammatory properties. J Periodontol. 2007 Apr;78(4):661-9. doi: 10.1902/jop.2007.060302. PMID 17397313
- [Background] Cieslik-Bielecka A, Gazdzik TS, Bielecki TM, Cieslik T. Why the platelet-rich gel has antimicrobial activity? Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Mar;103(3):303-5; author reply 305-6. doi: 10.1016/j.tripleo.2006.08.034. Epub 2007 Jan 2. No abstract available. PMID 17197209
- [Background] Filardo G, Kon E, Di Matteo B, Di Martino A, Tesei G, Pelotti P, Cenacchi A, Marcacci M. Platelet-rich plasma injections for the treatment of refractory Achilles tendinopathy: results at 4 years. Blood Transfus. 2014 Oct;12(4):533-40. doi: 10.2450/2014.0289-13. Epub 2014 Jun 19. PMID 24960641
- [Background] Dohan Ehrenfest DM, Andia I, Zumstein MA, Zhang CQ, Pinto NR, Bielecki T. Classification of platelet concentrates (Platelet-Rich Plasma-PRP, Platelet-Rich Fibrin-PRF) for topical and infiltrative use in orthopedic and sports medicine: current consensus, clinical implications and perspectives. Muscles Ligaments Tendons J. 2014 May 8;4(1):3-9. eCollection 2014 Jan. PMID 24932440
- [Background] Baksh N, Hannon CP, Murawski CD, Smyth NA, Kennedy JG. Platelet-rich plasma in tendon models: a systematic review of basic science literature. Arthroscopy. 2013 Mar;29(3):596-607. doi: 10.1016/j.arthro.2012.10.025. Epub 2013 Jan 24. PMID 23352397
- [Background] Mazzocca AD, McCarthy MB, Chowaniec DM, Dugdale EM, Hansen D, Cote MP, Bradley JP, Romeo AA, Arciero RA, Beitzel K. The positive effects of different platelet-rich plasma methods on human muscle, bone, and tendon cells. Am J Sports Med. 2012 Aug;40(8):1742-9. doi: 10.1177/0363546512452713. Epub 2012 Jul 16. PMID 22802273
- [Background] Gosens T, Peerbooms JC, van Laar W, den Oudsten BL. Ongoing positive effect of platelet-rich plasma versus corticosteroid injection in lateral epicondylitis: a double-blind randomized controlled trial with 2-year follow-up. Am J Sports Med. 2011 Jun;39(6):1200-8. doi: 10.1177/0363546510397173. Epub 2011 Mar 21. PMID 21422467
- [Derived] Walecka J, Bakowski P, Jokiel M, Trabka R, Chaszczewska-Markowska M, Ghete D, Gurda-Wozna D, Fedoruk-Wyszomirska A, Lubiatowski P, Wyszko E, Tyczewska A, Bakowska-Zywicka K. Molecular background behind lateral elbow pain reduction with Leukocyte-Rich and Leukocyte-Poor Platelet-Rich Plasma-randomized control trial and single-cell platelet analysis. Int Orthop. 2026 Jan 24. doi: 10.1007/s00264-025-06719-6. Online ahead of print. PMID 41579194